CLINICAL TRIAL: NCT03714776
Title: A Double-Blind, Placebo-Controlled, Phase 2 Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx, an Antisense Inhibitor Administered Subcutaneously to Hypertensive Subjects With Controlled Blood Pressure
Brief Title: A Study to Assess the Safety, Tolerability and Efficacy of IONIS-AGT-LRx, an Antisense Inhibitor Administered Subcutaneously to Hypertensive Participants With Controlled Blood Pressure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ISIS 757456-CS2
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Results first posted 2023-01-06 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2022-12

CONDITIONS: Mild Hypertension
Keywords: Hypertension; Hypertensive; AGT; Angiotensinogen; Blood Pressure; High Blood Pressure
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo matching solution injected subcutaneously (SC) once weekly for up to 6 weeks and an additional loading dose on Day 3.
  Interventions: Drug: Placebo
- ISIS 757456 80 mg (Experimental): ISIS 757456 80 mg injected SC once weekly for up to 6 weeks and an additional loading dose of 80 mg on Day 3.
  Interventions: Drug: ISIS 757456

INTERVENTIONS:
Drug: Placebo — Placebo matching solution administered as SC injection.
  Arms: Placebo
Drug: ISIS 757456 — Administered as SC injection.
  Other Names: IONIS-AGT-LRx
  Arms: ISIS 757456 80 mg

SUMMARY:
This was a Phase 2, double-blind, randomized, placebo-controlled study of IONIS-AGT-LRx conducted in mild hypertensive participants.

DETAILED DESCRIPTION:
Participants were randomized in a 2:1 ratio to receive a once-weekly subcutaneous treatment and an additional loading dose on Study Day 3 with either IONIS-AGT-LRx or placebo for 6 weeks.

All participants completed a 13-week Post-Treatment Period.

ELIGIBILITY:
Inclusion Criteria

1. Females must be non-pregnant and non-lactating, and either surgically sterile or post-menopausal.
2. Males must be surgically sterile or, abstinent or, if engaged in sexual relations with a woman of child-bearing potential, the participant or the participant's non-pregnant female partner must be using a highly effective contraceptive method
3. Body Mass Index (BMI) ≤ 35.0 kg/m2
4. Participant must have been diagnosed with essential hypertension for a minimum of 3 months prior to screening
5. At Screening, on a stable regimen of antihypertensive medications for at least 1 month prior to screening
6. Agree to conduct at home Blood Pressure (BP) and Heart Rate (HR) monitoring three times weekly and document the average of the triplicate measurements assessed on a day in the patient diary

Exclusion Criteria

1. Clinically-significant (CS) abnormalities in medical history, screening laboratory results, physical or physical examination that would render a participant unsuitable for inclusion
2. The use of the following at time of screening and during the course of the study:

   1. Other medications for the treatment of hypertension (e.g., clonidine, guanfacine, guanabenz, alpha-methyldopa, hydralazine, minoxidil, diazoxide, renin inhibitors)
   2. Medications that also may cause hyperkalemia (e.g., cyclosporine or tacrolimus, pentamidine, trimethoprim-sulfamethoxazole, all heparins)
   3. Oral or subcutaneous anticoagulants (e.g., warfarin, rivaroxaban, apixaban, heparin, lovenox)
   4. Organic nitrate preparations (e.g., nitroglycerin, isosorbide mononitrate, isosorbide dinitrate, or pentaerythritol)
   5. Sildenafil, tadalafil, vardenafil
3. Unwilling to discontinue antihypertensive mediations during Wash Out (WO) and Treatment Period of study
4. Participant has a history of secondary hypertension
5. Unstable/underlying cardiovascular disease defined as:

   1. Any history of congestive heart failure (NYHA class II-IV)
   2. Any history of previous stroke, transient ischemic attack, unstable or stable angina pectoris, or myocardial infarction prior to screening
   3. a history or evidence of long QT syndrome
   4. Any CS active atrial or ventricular arrhythmias
   5. Any history of coronary bypass or percutaneous coronary intervention

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Orange County Research Center, Tustin, California
  - Progressive Medical Research, Port Orange, Florida
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - Ohio Clinical Research - Lyndhurst, Lyndhurst, Ohio
  - Juno Research, LLC - Northwest Site, Houston, Texas
  - York Clinical Research LLC, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in the United States from 03 January 2019 to 13 November 2019.
Pre-assignment Details: A total of 77 participants were screened of which 25 were enrolled and randomized to receive study drug.
Period: Overall Study
Arm/Group | Placebo | ISIS 757456 80 mg
Started | 8 | 17
Safety Set (Safety Set included all participants who were randomized and received at least 1 dose of study drug.) | 8 | 17
Full Analysis Set (FAS) (FAS included all randomized participants who received at least 1 injection of study drug and who had at least 1 post-Baseline efficacy or exploratory measurements.) | 8 | 17
Per Protocol Set (PPS) (PPS included all FAS participants who received at least 5 of the 7 doses of study drug, did not receive antihypertensive medications during the Treatment Period and prior to Day 43, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.) | 6 | 15
Completed | 8 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who were randomized and received at least 1 dose of study drug.
Groups:
- Placebo: Placebo matching solution injected SC once weekly for up to 6 weeks and an additional loading dose on Day 3.
- Total: Total of all reporting groups
Arm/Group | Placebo | ISIS 757456 80 mg | Total
Number analyzed (Participants) | 8 | 17 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (4) | 60 (7) | 59 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 2 | 10 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 10
  Not Hispanic or Latino | 6 | 9 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 5 | 10 | 15
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Plasma Angiotensinogen (AGT) Concentration [Mean (Full Range); unit: micrograms per milliliter (μg/mL)] — Population: PPS: All FAS(all randomized participants who received at least 1 injection of study drug and who had at least 1 post-Baseline efficacy or exploratory measurements) participants who received at least 5 of the 7 doses of study drug, did not receive antihypertensive medications during Treatment Period and prior to Day 43, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.
  micrograms per milliliter (μg/mL)
    number analyzed (Participants) | 6 | 15 | 21
    (all) | 19.5 [15.4 to 25.4] | 20.3 [14.1 to 28.3] | 19.9 [14.1 to 28.3]
In-clinic Systolic Blood Pressure (SBP) [Mean (Full Range); unit: millimeters of mercury (mmHg)] — Population: PPS: All FAS (all randomized participants who received at least 1 injection of study drug and who had at least 1 post-Baseline efficacy or exploratory measurements) participants who received at least 5 of the 7 doses of study drug, did not receive antihypertensive medications during Treatment Period and prior to Day 43, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.
  millimeters of mercury (mmHg)
    number analyzed (Participants) | 6 | 15 | 21
    (all) | 148 [128 to 163] | 145 [133 to 167] | 145.9 [128 to 167]

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Plasma Angiotensinogen (AGT) at Day 43 (Week 7) Compared to Placebo
Time Frame: Baseline, Week 7
Population: PPS included all FAS participants (all randomized participants who received at least 1 injection of study drug and who had at least 1 post-Baseline efficacy or exploratory measurements) who received at least 5 of the 7 doses of the study drug, did not receive antihypertensive medications during the Treatment Period and prior to Day 43, and had no significant protocol deviations that would have been expected to affect efficacy or exploratory assessments.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ISIS 757456 80 mg
Number analyzed (Participants) | 6 | 15
percent change | 12.6 (23.3) | -54.2 (24.8)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456 80 mg; Test type: Superiority; p < 0.001, ANOVA — P-value of analysis of variance (ANOVA) with treatment and screening AGT concentration stratification factor was used for analysis

2. Secondary Outcome: Change From Baseline in the In-clinic Systolic Blood Pressure (SBP) at Days 3, 8, 15, 22, 29, and 36
Time Frame: Baseline, Days 3, 8, 15, 22, 29, and 36
Population: PPS=all FAS participants(all randomized participants who received at least 1 injection of study drug and had at least 1 post-Baseline efficacy or exploratory measurements)who received at least 5 of 7 doses of study drug, did not receive antihypertensive medications during Treatment Period prior to Day 43, had no significant protocol deviations that would have been expected to affect efficacy assessments. Number analyzed=number of participants with data available for analysis at given time point.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | ISIS 757456 80 mg
Number analyzed (Participants) | 6 | 15
mmHg
  Change From Baseline at Day 3 | -10 (4) | -7 (10)
  Change From Baseline at Day 8 | -6 (18) | -5 (12)
  Change From Baseline at Day 15: number analyzed (Participants) | 6 | 14
  Change From Baseline at Day 15 | -14 (10) | -4 (14)
  Change From Baseline at Day 22 | -10 (12) | -7 (14)
  Change From Baseline at Day 29 | -1 (13) | -5 (11)
  Change From Baseline at Day 36 | -3 (10) | -8 (13)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456 80 mg; Day 3; Test type: Superiority; p = 0.454, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 2: Comparison: Placebo vs ISIS 757456 80 mg; Day 8; Test type: Superiority; p = 0.909, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 3: Comparison: Placebo vs ISIS 757456 80 mg; Day 15; Test type: Superiority; p = 0.132, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 4: Comparison: Placebo vs ISIS 757456 80 mg; Day 22; Test type: Superiority; p = 0.659, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 5: Comparison: Placebo vs ISIS 757456 80 mg; Day 29; Test type: Superiority; p = 0.474, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 6: Comparison: Placebo vs ISIS 757456 80 mg; Day 36; Test type: Superiority; p = 0.483, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis

3. Secondary Outcome: Percent Change From Baseline in Plasma AGT at Days 3, 8, 15, 22, 29 and 36
Time Frame: Baseline, Days 3, 8, 15, 22, 29, and 36
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | ISIS 757456 80 mg
Number analyzed (Participants) | 6 | 15
percent change
  Percent Change From Baseline at Day 3 | 6.8 (20.5) | -8.3 (13.8)
  Percent Change From Baseline at Day 8 | 19.1 (23.8) | -35.7 (13.8)
  Percent Change From Baseline at Day 15: number analyzed (Participants) | 6 | 14
  Percent Change From Baseline at Day 15 | 7.6 (28.2) | -50.4 (16.4)
  Percent Change From Baseline at Day 22 | 8.7 (24.0) | -52.4 (17.3)
  Percent Change From Baseline at Day 29 | 6.1 (13.8) | -62.2 (10.5)
  Percent Change From Baseline at Day 36 | 2.9 (27.7) | -58.3 (12.9)
Statistical Analysis 1: Comparison: Placebo vs ISIS 757456 80 mg; Day 3; Test type: Superiority; p = 0.064, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 2: Comparison: Placebo vs ISIS 757456 80 mg; Day 8; Test type: Superiority; p < 0.001, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 3: Comparison: Placebo vs ISIS 757456 80 mg; Day 15; Test type: Superiority; p < 0.001, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 4: Comparison: Placebo vs ISIS 757456 80 mg; Day 22; Test type: Superiority; p < 0.001, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 5: Comparison: Placebo vs ISIS 757456 80 mg; Day 29; Test type: Superiority; p < 0.001, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis
Statistical Analysis 6: Comparison: Placebo vs ISIS 757456 80 mg; Day 36; Test type: Superiority; p < 0.001, ANOVA — P-value of ANOVA with treatment and screening AGT concentration stratification factor was used for analysis

ADVERSE EVENTS:
Time Frame: Up to Week 19
Description: Safety Set included all participants who were randomized and received at least 1 dose of study drug.
Arm/Group | Placebo | ISIS 757456 80 mg
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/17
Other Adverse Events (participants affected / at risk) | 7/8 | 8/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | ISIS 757456 80 mg (N=17)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8) | ISIS 757456 80 mg (N=17)
Injection site erythema (General disorders) | 0 | 2
Chills (General disorders) | 1 | 0
Injection site haemorrhage (General disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 1
Injection site swelling (General disorders) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 2 | 0
Headache (Nervous system disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT03714776/Prot_SAP_001.pdf